CLINICAL TRIAL: NCT02015507
Title: An Open-Label, Phase 1 Study in Healthy Adult Subjects to Examine the Effects of Multiple-Dose Ciprofloxacin on the Multiple-Dose Pharmacokinetics of Ivacaftor and on the Multiple-Dose Pharmacokinetics of VX-661 Administered in Combination With Ivacaftor
Brief Title: An Open-Label, Phase 1 Study in Healthy Adult Subjects to Examine the Effects of Multiple-Dose Ciprofloxacin on Ivacaftor and VX-661 in Combination With Ivacaftor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VX13-770-017
Record Dates: First submitted 2013-12-09; First posted 2013-12-19 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor; tezacaftor; Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Active Comparator): participants in Cohort 1 will be administered ivacaftor alone followed by ivacaftor with concomitant ciprofloxacin.
  Interventions: Drug: ivacaftor; Drug: ciprofloxacin
- Cohort 2 (Experimental): Participants in Cohort 2 will be administered VX-661 in combination with ivacaftor followed by VX-661 in combination with ivacaftor and concomitant ciprofloxacin
  Interventions: Drug: ivacaftor; Drug: VX-661; Drug: ciprofloxacin

INTERVENTIONS:
Drug: ivacaftor
Drug: VX-661
  Arms: Cohort 2
Drug: ciprofloxacin

SUMMARY:
To evaluate the effect of ciprofloxacin on the pharmacokinetics (PK) of ivacaftor and on the pharmacokinetics of VX-661 when administered in combination with ivacaftor

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with scheduled visits, treatment plan, study restrictions,laboratory tests, contraception guidelines, and other study procedures
* Healthy subjects, as defined by no clinically relevant abnormalities identified by a detailed medical history and full physical examination, including blood pressure and heart rate measurement, standard 12-lead ECG, and clinical laboratory tests.
* Body mass index (BMI) of 18.0 to 31.0 kg/m2, inclusive, and a total body weight >50 kg
* Female subjects of childbearing potential must have a negative serum pregnancy test at screening and at the Day -1 Visit.

Exclusion Criteria:

* History of any illness, clinical condition, or other factor that, in the opinion of the investigator or the subject's general practitioner, might confound the results of the study or pose an additional risk in administering study drug(s) to the subject
* Inability to swallow capsules, or inadequate venous access.
* History of febrile illness within 5 days before the first study drug dose
* A screen positive for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus 1 or 2 antibodies.
* For female subjects: Pregnant or nursing subjects and female subjects of childbearing potential who are unwilling or unable to use an acceptable method of contraception as outlined in this protocol. For male subjects: Subject has a female partner who is pregnant, nursing, or planning to become pregnant during the study or within 120 days after the last study drug dose.
* Any condition possibly affecting drug absorption
* Abnormal renal function at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
PK parameters of ivacaftor and metabolites following concomitant dosing with ciprofloxacin relative to ivacaftor administered alone | Day 7, Day 14
  PK Parameters - maximum observed plasma concentrations (Cmax) and area under the concentration versus time curve (AUC),
PK parameters of VX-661 and metabolites when dosed in combination with ivacaftor and concomitant ciprofloxacin relative to VX-661 administered in combination with ivacaftor | Day 10, Day 20
  PK parameters - maximum observed plasma concentrations (Cmax) and area under the concentration versus time curve (AUC),

SECONDARY OUTCOMES:
PK parameters of ivacaftor and metabolites when administered in combination with VX-661, with and without concomitant ciprofloxacin | Day 10, Day 20
  PK Parameters - maximum observed plasma concentrations (Cmax) and area under the concentration versus time curve (AUC),
Safety and tolerability, as assessed by adverse events (AEs), vital signs, ECGs and laboratory assessments | Day 1 through Day 21 (cohort 1) or Day 34 (cohort2)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceutical Incorporated